CLINICAL TRIAL: NCT00867373
Title: Parent Perceptions of Weight Status: Impact of a Pilot Intervention to Enhance Awareness of Risk for Overweight Parents and Their Children
Brief Title: Parent Perceptions of Weight Status: Impact of a Pilot Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 07-0329
Record Dates: First submitted 2009-03-19; First posted 2009-03-23 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
Keywords: Obesity; Weight perceptions
MeSH Terms: conditions — Obesity | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education Intervention (Experimental): The intervention used in the randomized controlled trial consists of 1) measuring the parents' height and weight and 2) providing the parents with feedback on their calculated BMI on an educational handout (included in Appendix V). The purpose of the handout is to convey the following 5 messages:
  1. Definition of BMI
  2. How BMI is calculated
  3. What the parent's BMI is based on the measurements taken
  4. What weight category the parent is in (underweight, normal weight, overweight, or obese)
  5. Children with overweight or obese parents are at higher risk of becoming overweight themselves.
  The Research Assistant will verbally review the educational handout with the parent. The handout will be available in both English and Spanish.
  Interventions: Behavioral: Education Intervention
- Control Group (No Intervention): Parents assigned to the control group will proceed to their child's well child visit after their baseline data are collected.

INTERVENTIONS:
Behavioral: Education Intervention — The intervention is a short educational handout regarding BMI and the effect of parental weight status on children.
  Arms: Education Intervention

SUMMARY:
This pilot study is a randomized controlled trial with an embedded cross sectional study exploring parental perceptions of their weight status and how it affects their perceptions of their child's weight status. This study uses an educational intervention in which parents are informed of their actual weight status and how it affects their child's health. We will study the effect of this intervention on the parent's perceptions of and level of concern for their own and their child's weight status.

DETAILED DESCRIPTION:
Pediatric obesity has tripled in the past 20 years. Obesity prevention early in life is important and parental participation is essential. Parents must recognize overweight in their child so health providers may engage them in a dialogue to change their child's diet and physical activity patterns, yet a large proportion of parents do not recognize that their child is overweight. Parents' misperception of their overweight child's weight status presents a barrier to treating obesity.

This pilot study is a randomized controlled trial with an embedded cross sectional study exploring parental perceptions of their weight status and how it affects their perceptions of their child's weight status. This study uses an educational intervention in which parents are informed of their actual weight status and how it affects their child's health. We will study the effect of this intervention on the parent's perceptions of and level of concern for their own and their child's weight status.

Our goal is to develop a primary care intervention that will enhance parental perceptions of overweight and motivation to make changes for their family. Pilot data collected here will support an R21 Exploratory/Developmental Clinical Research Grant in Obesity or a Centers for Disease Control (CDC) or Robert Wood Johnson Foundation (RWJ) grant submission.

ELIGIBILITY:
Inclusion Criteria:

1. Boys and girls ages 3 to 13 years old presenting with at least one biological parent for a routine health maintenance exam (WCC) at the Child Health Continuity Clinic will be eligible. Parents must be able and willing to have their height and weight measured at the clinic

Exclusion Criteria:

1. Child has previously been referred to a nutritionist/dietician or specialized clinic/program for weight management
2. Child is currently being treated for failure to thrive
3. Child is on parenteral nutrition
4. Child is on chronic systemic steroid therapy
5. Child is non-mobile/wheelchair bound
6. The family has previously enrolled into the study with a prior sibling
7. Family is unable to be contacted at home
8. Presenting parent cannot speak and read English or Spanish at at least a 5th grade level

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Proportion of parents correctly assessing their own weight status | At first visit

SECONDARY OUTCOMES:
Proportion of parents correctly assessing their child's weight status | At first visit
Proportion of parents who underestimate own weight status who also underestimate their child's weight status | At first visit
Change in proportion of parents underestimating their own weight status | At first visit and at one week follow up phone survey
Change in proportion of parents underestimating their child's weight status | At first visit and at one week follow up phone survey
Change in level of concern pre- and post-intervention | At first visit and at one week follow up phone survey

CONTACTS AND LOCATIONS:
Overall Officials: Christina Suh, MD, Principal Investigator — University of Colorado, Denver; Nancy F. Krebs, MD, Principal Investigator — University of Colorado, Denver; Allison Kempe, MD, MPH, Principal Investigator — Univeristy of Colorado Denver
Locations (1):
- The Children's Hospital, Aurora, Colorado, United States

REFERENCES:
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Daniels SR, Arnett DK, Eckel RH, Gidding SS, Hayman LL, Kumanyika S, Robinson TN, Scott BJ, St Jeor S, Williams CL. Overweight in children and adolescents: pathophysiology, consequences, prevention, and treatment. Circulation. 2005 Apr 19;111(15):1999-2012. doi: 10.1161/01.CIR.0000161369.71722.10. PMID 15837955
- [Background] Rhee KE, De Lago CW, Arscott-Mills T, Mehta SD, Davis RK. Factors associated with parental readiness to make changes for overweight children. Pediatrics. 2005 Jul;116(1):e94-101. doi: 10.1542/peds.2004-2479. PMID 15995022
- [Background] Logue E, Sutton K, Jarjoura D, Smucker W. Obesity management in primary care: assessment of readiness to change among 284 family practice patients. J Am Board Fam Pract. 2000 May-Jun;13(3):164-71. doi: 10.3122/15572625-13-3-164. PMID 10826863
- [Background] Wee CC, Davis RB, Phillips RS. Stage of readiness to control weight and adopt weight control behaviors in primary care. J Gen Intern Med. 2005 May;20(5):410-5. doi: 10.1111/j.1525-1497.2005.0074.x. PMID 15963162
- [Background] Eckstein KC, Mikhail LM, Ariza AJ, Thomson JS, Millard SC, Binns HJ; Pediatric Practice Research Group. Parents' perceptions of their child's weight and health. Pediatrics. 2006 Mar;117(3):681-90. doi: 10.1542/peds.2005-0910. PMID 16510647
- [Background] Jeffery AN, Voss LD, Metcalf BS, Alba S, Wilkin TJ. Parents' awareness of overweight in themselves and their children: cross sectional study within a cohort (EarlyBird 21). BMJ. 2005 Jan 1;330(7481):23-4. doi: 10.1136/bmj.38315.451539.F7. Epub 2004 Nov 26. No abstract available. PMID 15567804
- [Background] Birch LL, Fisher JO. Development of eating behaviors among children and adolescents. Pediatrics. 1998 Mar;101(3 Pt 2):539-49. PMID 12224660
- [Background] Epstein LH, Wing RR, Koeske R, Andrasik F, Ossip DJ. Child and parent weight loss in family-based behavior modification programs. J Consult Clin Psychol. 1981 Oct;49(5):674-85. doi: 10.1037//0022-006x.49.5.674. No abstract available. PMID 7287977
- [Background] Golan M, Weizman A, Apter A, Fainaru M. Parents as the exclusive agents of change in the treatment of childhood obesity. Am J Clin Nutr. 1998 Jun;67(6):1130-5. doi: 10.1093/ajcn/67.6.1130. PMID 9625084